CLINICAL TRIAL: NCT06899321
Title: A Clinical Study to Evaluate Test Products for Skin Brightening Benefit Under Controlled UV Exposure, in a 6-week Study Design
Brief Title: The Effect of Cosmetic Products on Skin Brightening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: MS Clinical Research Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SKN-SKA-4328
Record Dates: First submitted 2025-03-11; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Skin Brightening

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will receive all study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cosmetic product M68 (Experimental): Cosmetic product to be applied twice daily 6 days a week (except on measurement days, when it will be applied once) for the duration of the study.
  Interventions: Other: Cosmetic product M68
- Cosmetic product Z15 (Experimental): Cosmetic product to be applied twice daily 6 days a week (except on measurement days, when it will be applied once) for the duration of the study.
  Interventions: Other: Cosmetic product Z15
- Cosmetic product R52 (Experimental): Cosmetic product to be applied twice daily 6 days a week (except on measurement days, when it will be applied once) for the duration of the study.
  Interventions: Other: Cosmetic product R52
- Cosmetic product J61 (Experimental): Cosmetic product to be applied twice daily 6 days a week (except on measurement days, when it will be applied once) for the duration of the study.
  Interventions: Other: Cosmetic product J61
- Cosmetic product U36 (Experimental): Cosmetic product to be applied twice daily 6 days a week (except on measurement days, when it will be applied once) for the duration of the study.
  Interventions: Other: Cosmetic product U36
- No treatment control (No Intervention): No treatment control

INTERVENTIONS:
Other: Cosmetic product M68 — Cosmetic skin brightening product to be applied to defined test site
  Arms: Cosmetic product M68
Other: Cosmetic product Z15 — Cosmetic skin brightening product to be applied to defined test site
  Arms: Cosmetic product Z15
Other: Cosmetic product R52 — Cosmetic skin brightening product to be applied to defined test site
  Arms: Cosmetic product R52
Other: Cosmetic product J61 — Cosmetic skin brightening product to be applied to defined test site
  Arms: Cosmetic product J61
Other: Cosmetic product U36 — Cosmetic skin brightening product to be applied to defined test site
  Arms: Cosmetic product U36

SUMMARY:
This is a single centre, single cell, blinded study designed to evaluate the effect of 5 cosmetic products on skin brightening, skin hydration and skin barrier function of the volar forearm after controlled UV exposure as compared to baseline and a no-treatment control.

DETAILED DESCRIPTION:
This is a single centre, single cell, blinded study designed to evaluate the effect of cosmetic products on skin brightening, skin hydration and skin barrier function of the volar forearm after controlled UV exposure. This study will accept 34 participants who meet the inclusion and exclusion criteria. Participants will test all 5 products and a no-treatment control, which will be applied twice daily for 6 weeks to pre-defined test sites on their volar forearms.

UV exposure will be conducted using a SOL UV solar simulator (300 - 1200nm; dose level 6 joules/cm2) at various time points during weeks 2 - 5 of the study.

Instrumental assessments of skin brightening, skin hydration and skin barrier function will be conducted at regular intervals throughout the whole study. Non-invasive samples of the stratum corneum will be collected at several timepoints during the study to evaluate biomarkers of skin brightening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female adult participants in general good health as determined from a recent medical history.
* Participants in the age group of 18-45 years as on the day of enrolment (both ages inclusive).
* Participants having very little hair, no burns, no cut/abrasion; no moles/tattoo/birth marks/burn marks on the test sites/areas as identified on screening.
* Participants with long and broad forearms.
* Participants having skin photo-type IV and V.
* Participants with Spectrophotometer L* value- 45 to 55 (both values included) on the identified test sites on the volar forearm.
* Participants having uniform skin color and no sunburn/ erythema on the test sites.
* Participants who do not have very dry or scaly skin, uneven skin tone on their volar forearms or no other signs of significant local irritation or skin disease like psoriasis.
* Participants who agree to refrain from using pumice stone, scrubber while bathing during the study.
* Participants who are willing to avoid direct sun exposure to the test sites.
* Participants who have not participated in any clinical product evaluation test within past 1 month.
* Participants able to read and sign an appropriate informed consent form indicating her willingness to participate and agree to come for regular study visits.
* Participants willing to abide by and comply with the study protocol.
* Participants willing to use umbrella & wear full covered attire if she has to go in sun.
* Participants who are willing not to participate in any other clinical study during participation in the current study.

Exclusion Criteria:

* Participants with a known history or present condition of allergic response to any sunscreen products, cosmetic products, bathing soaps, detergent powder or medicine.
* Participants who have outdoor job, extremely physical (manual) job which could cause excessive sun exposure or sweating
* Participants who are smokers.
* Menopausal women.
* Participants having active skin diseases which will interfere with the test readings.
* Participants on oral and topical medications (e.g Steroids, anti-oxidant, antibiotics) which will compromise the study.
* Systemic treatment which may modify the cutaneous state on the day of inclusion or in the previous 30 days, including retinoid therapy.
* Participants who are pregnant, lactating or nursing.
* Intense sun exposure/ photo allergenicity/toxicity.
* Chronic illness which may influence the cutaneous state.
* Participants participating in any other cosmetic or therapeutic trial.
* Participants with any underlying uncontrolled medical illness including diabetes mellitus, hypertension, liver disease or history of alcoholism, HIV, hepatitis, or any other serious medical illness that will pose a health risk due to study participation as per investigator's discretion.
* For female participants only: be pregnant, planning pregnancy or lactating/nursing. Urine pregnancy testing (UPT) will be performed at the time of screening.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
L* measured using CM2600D | 0 - 6 weeks
  L* (Luminance) - represents lightness/darkness values of luminosity indices (total quantity of light reflected). L* is measured using spectrophotometer CM2600D, which measures the spectral reflectance in the visible wavelength range of 400nm to 700nm as the ratio of the power of the net total reflected light over total incident light. The colour values of L*a*b* are calculated from the spectral reflectance.
  * Manufacturer Name: Konica Minolta
  * Measurement Range: L* 0 - 100
  * Efficacy Direction of L*: Higher is better

SECONDARY OUTCOMES:
a* measured using CM2600D | 0 - 6 weeks
  a* (Red/green component of CIELAB colour space). a* represents colour ranging from red to green - positive values are red; negative values are green.
  a* is measured using a spectrophotometer CM2600D, which measures the spectral reflectance in the visible wavelength range of 400nm to 700nm as the ratio of the power of the net total reflected light over total incident light. The colour values of L*a*b* are calculated from the spectral reflectance.
  * Manufacturer Name: Konica Minolta
  * Measurement Range: a* -128 to 127
  * Efficacy Direction of a*: +a is redder, -a is greener
Skin hydration measured using Corneometer CM825 | 0 - 6 weeks
  The corneometer (CM825) indirectly measures the skin's hydration as a change in capacitance of the stratum corneum.
  * Manufacturer Name: MPA (Multiprobe Adaptor) unit from C&K (Courage & Khazaka)
  * Depth of measurement approximately 45 μm
  * Measurement Range: 0 - 120 Arbitrary Units (AU)
  * Efficacy Direction of Corneometer reading: Higher is better
Skin barrier function (Trans-Epidermal Water Loss [TEWL]) measured using Tewameter TM300 | 0 - 6 weeks
  Skin barrier function (TEWL) is measured using the Tewameter TM300.
  * Manufacturer Name: MPA (Multiprobe Adaptor) unit from C&K (Courage Khazaka)
  * Measurement Range: 0 - 250 g/m²/h
  * Efficacy Direction of TEWL reading: Lower is better

OTHER OUTCOMES:
Stratum corneum biomarkers of skin brightening | 0 - 6 weeks
  Biomarkers associated with skin brightening will be measured from non-invasive D-Squame tape-strip samples of the stratum corneum.
  Up to 15 sequential tape strips will be collected.
  The following biomarkers will be analysed using ELISA:
  Filaggrin: measure of skin barrier. ng/ml. Efficacy: higher is better. IL1a: measure of inflammation. pg/ml. Efficacy: lower is better. IL1RA: measure of inflammation. pg/ml. Efficacy: lower is better. Catalase: measure of antioxidant effect. pg/ml. Efficacy: higher is better. Total antioxidant. mmol/L. Efficacy: higher is better.
  Total protein will also be measured.
  Additional biomarkers related to the objectives may also be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- MS Clinical Research Pvt Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No